CLINICAL TRIAL: NCT06847074
Title: Rise & Shine: Promoting Sleep Quality in Chronic Stroke With Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H23-01163
Record Dates: First submitted 2025-02-17; First posted 2025-02-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Poor Quality Sleep
Keywords: Exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Exercise Training (Experimental): The program will consist of moderate intensity, multimodal exercise training; 2x/week; in-person, group-based.
  Interventions: Behavioral: Multimodal Exercise
- Cognitive and Social Activities (No Exercise) (Active Comparator): The program will consist of cognitive and social activites; 2x/week; in-person, group-based
  Interventions: Behavioral: Cognitve and Social Activities

INTERVENTIONS:
Behavioral: Multimodal Exercise — Each 60-minute class will include a 10-minute warm-up (i.e., stretches for the major muscles and walking on the spot), 40 minutes of training, and a 10-minute cool down (i.e., stretches and relaxation techniques).Instructors will use heart rate monitors to continuously track intensity during and across all sessions.
  Arms: Multimodal Exercise Training
Behavioral: Cognitve and Social Activities — Each 60-minute class will include 30 minutes of cognitive enrichment activities and 30 minutes of activities that promote social interactions.
  Arms: Cognitive and Social Activities (No Exercise)

SUMMARY:
health problems, such as heart disease, diabetes, cognitive impairment, and dementia.

After a person suffers a stroke, they often experience difficulties in getting a good night's sleep. Approximately half of stroke survivors have insomnia, or have trouble falling and/or staying asleep. Poor sleep quality among stroke survivors increases the risk of recurrent stroke by 3-fold and the risk of early death by 76%. Hence, stroke survivors need strategies to promote better sleep.

Fortunately, evidence shows that sleep quality can be improved with exercise, even among those who struggle with insomnia. Whether exercise training can improve sleep quality in adults with chronic stroke (i.e., at least 12 months has passed since their stroke) and poor sleep quality is not known. In addition, it is unknown if improved sleep is associated with improved outcomes in those with chronic stroke.

This study will specifically evaluate the effect of twice-weekly targeted exercise training on sleep quality over a 6-month period in persons with chronic stroke and poor sleep quality. This study will also evaluate the effect of exercise on the following outcomes: 1) sleep structure; 2) fatigue; 3) daytime sleepiness; 4) mood; 5) physical function and capacity; 6) thinking abilities; 7) heart health; and 8) quality of life. Finally, this study will examine how changes in sleep quality may be related to changes in these outcomes. Our proposed research is timely as the importance of sleep to recovery, health, and wellbeing post-stroke is increasingly recognized.

DETAILED DESCRIPTION:
Approximately half of stroke survivors have insomnia. Poor sleep quality among stroke survivors increases the risk of recurrent stroke by 3-fold and the risk of early death by 76%. Hence, stroke survivors are a target population in need of intervention strategies to promote sleep quality.

Current research and stroke rehabilitation do not address the sleep consequences of stroke - especially for those in the chronic phase (i.e., = or > 12 months since an index stroke). Adults with chronic stroke have lower sleep efficiency compared with sex- and age-matched controls. Poor sleep quality in chronic stroke is associated with depression, impaired physical function, and reduced cognitive function.

How to effectively treat insomnia in adults with chronic stroke is not well established. Intervention studies show exercise improves sleep quality and structure. Whether exercise can improve sleep quality in adults with chronic stroke and poor sleep quality is not established.

Primary Question: In adults with chronic stroke and poor sleep quality, can a 26-week multimodal exercise training program of moderate intensity (EX) improve sleep efficiency, as objectively measured by the actigraphy, compared with a 26-week cognitive and social activities program (CON; active control group)?

Secondary Question: What are additional benefits of EX vs. CON? Compared with CON, we will evaluate the effect of EX on: 1) actigraphy-measured sleep parameters of latency, duration, and wake after sleep onset; 2) sleep architecture by frontal electroencephalography; 3) subjective sleep quality; 4) fatigue; 5) daytime sleepiness; 6) mood; 7) functional capacity; 8) cognitive function; 9) cardiometabolic risk factors; and 10) quality of life.

Tertiary Question: Are changes in sleep quality associated with changes in: 1) fatigue; 2) daytime sleepiness; 3) mood; 4) cognitive function; 5) cardiometabolic risk factors; and 6) quality of life?

Pilot Data: Using actigraphy, the investigators acquired sleep data from 21 of 120 (i.e., subset) participants with chronic stroke enrolled in a RCT with cognitive function as the primary outcome. These 21 participants (mean age=69) were randomized to 26 weeks of: 1) multimodal exercise of moderate intensity (EX; n=12); or 2) cognitive and social activities (i.e., no exercise; CON; n=9). Of these 21 participants, 48% had a baseline actigraphy-measured sleep efficiency < 85%. Compared with CON, EX significantly improved actigraphy-measured sleep efficiency values (in %) at 13 weeks and 26 weeks.

Methods: A 26-week, assessor-blinded, single-site RCT of 62 community-dwelling adults with chronic stroke, WatchPAT measured sleep efficiency < 85%, Pittsburgh Sleep Quality Index global score > 5, and aged 55 years and older. Individuals will be randomized to one of two experimental groups: 1) twice-weekly EX (n=31); or 2) twice-weekly CON (n=31). Randomization will be stratified by sex and age. Measurement will occur at baseline, 13 weeks, and 26 weeks, unless otherwise stated.

ELIGIBILITY:
Inclusion Criteria:

We will include community-dwelling adults who had an ischemic or hemorrhagic stroke at least one year prior to study enrolment and have poor sleep quality - defined as a sleep efficiency of < 85% and a PSQI global score of > 5. Individuals must also meet these inclusion criteria: 1) aged 55 years and older; 2) a baseline MMSE score of = or > 22/30 and a MoCA score of = or > 19/30; 3) community-dwelling; 4) able to comply with scheduled assessments, classes, and other trial procedures; 5) read, write, and speak English with acceptable visual and auditory acuity; 6) not to start or stable (i.e., = or > 6 months) on a fixed dose of medication that impacts sleep (i.e., anti-arrhythmics, beta blockers, selective serotonin reuptake inhibitor, etc.) during the 26-week intervention period; 7) able to walk for a minimum of six metres with rest intervals with or without assistive devices; 8) based on interview, have an activity tolerance of 60 minutes with rest intervals; 9) not participating in any regular therapy or progressive exercise (e.g., treadmill or weight-lifting); and 10) able to safely engage in exercise as indicated by the PAR-Q+63 and written confirmation by family or study physicians.

Exclusion Criteria:

We will exclude individuals who: 1) are diagnosed with OSA and are not using CPAP or defined as potentially having undiagnosed OSA (AHI > 20) as a result of study screening; 2) have restless leg syndrome; 3) are diagnosed with dementia of any type; 4) are diagnosed with another type of neurodegenerative or neurological condition (e.g., Parkinson's disease); 5) are planning to participate, or already enrolled in, a clinical drug trial or exercise trial concurrent to this study; 6) are at high risk for cardiac complications during exercise and/or unable to self-regulate activity or to understand recommended activity level; 7) have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility, as determined by his/her physician; or 8) have aphasia as judged by an inability to communicate by phone.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | Baseline, 13 weeks, 26 weeks
  Sleep efficiency as measured by actigraphy over days of wear.

SECONDARY OUTCOMES:
Sleep latency, duration, and wake after sleep onset | Baseline, 13 weeks, 26 weeks
  Sleep latency, duration, and wake after sleep onset by actigraphy over days of wear.
Sleep architecture (OPTIONAL) | Baseline, 13 weeks, 26 weeks
  Sleep architecture as measured by EEG headband
Subjective sleep quality | Baseline, 13 weeks, 26 weeks
  Subjective sleep quality measured by Pittsburgh Sleep Quality Index
Fatigue | Baseline, 13 weeks, 26 weeks
  Fatigue measured by Fatigue Severity Scale
Sleepiness | Baseline, 13 weeks, 26 weeks
  Daytime sleepiness measured by questionnaire
Mood | Baseline, 13 weeks, 26 weeks
  Depressive symptoms measured by questionnaire
Functional capacity | Baseline, 13 weeks, 26 weeks
  Functional capacity, or aerobic capacity, measured by the 6-Minute Walk Test
NIH Toolbox Cognitive Battery | Baseline, 13 weeks, 26 weeks
  Cognitive function measured by NIH Toolbox Cognitive Battery
ADAS-Cog Plus | Baseline, 13 weeks, 26 weeks
  Cognitive function measured by ADAS-Cog Plus
Executive Functions | Baseline, 13 weeks, 26 weeks
  The domain of executive functions measured by Trails A and B, Digits Forward and Backward, and Clock Drawing
Verbal Fluency | Baseline, 13 weeks, 26 weeks
  Verbal fluency measured by categorical fluency
Memory | Baseline, 13 weeks, 26 weeks
  Memory measured by the Rey Auditory Verbal Fluency
Blood pressure | Baseline, 13 weeks, 26 weeks
  Systolic and diastolic blood pressure
Chronotype | Baseline, 13 weeks, 26 weeks
  Chronotype measured by questionnaire
Blood biomarkers (OPTIONAL) | Baseline, 13 weeks, 26 weeks
  We will draw blood to assess markers cardiometabolic health and brain health
Quality of life | every 4 weeks, up to 26 weeks
  Quality of Life measured by the EuroQol-5 Domain-5 Level (EQ-5D-5L)
Current physical activity | every 4 weeks, up to 26 weeks
  Physical activity outside of research study will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health Research Institute Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No